CLINICAL TRIAL: NCT04908540
Title: Evaluatin of Maxillery Skeletal Expansion in Young Adults, With Two Different Activation Protocols. A Randomized Clinical Trial
Brief Title: New Maxillary Expansion Technique in Adults
Acronym: ALT/MARPE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiti Sains Malaysia (Other)
Collaborators: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Amira Hussein Ahmed Mohamed Allam, Dr., Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PhD Amira USM
Record Dates: First submitted 2021-05-25; First posted 2021-06-01 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Maxillary Dysostosis (Disorder)
Keywords: Adult Maxillary Expansion; Activation Protocols

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MARPE/ Conventional (Control) (Group A) (Active Comparator): patients will open the appliance in its conventional way; 2 quarter turn (0.2 mm) in the morning, and 2 quarter turn in the evening until overcorrection achieved.
  Interventions: Procedure: Mini-screw Assissted Rapid Palatal Expansion
- MARPE/ ALT-RAMEC (Group B) (Experimental): Patients will open 2 quarter turn (0.2mm) in the morning, and 2 in the evening in the first week, then alternate with closing 2 quarter turn in the morning and 2 in the evening in the second week. And then continuing opening and closing till end with opening in the 7th week and continue opening until overcorrection achieved.
  Interventions: Procedure: Mini-screw Assissted Rapid Palatal Expansion

INTERVENTIONS:
Procedure: Mini-screw Assissted Rapid Palatal Expansion — Mini-screw assissted RPE will be the main intervention in the two comparative groups. In the control (group A) will be used with its conventional activation protocol. While in experimental (group B) will be used with ALT-RAMEC protocol.
  Other Names: Maxillary Skeletal Expansion

SUMMARY:
Previous studies confirmed that MARPE (Mini-screw Assisted Rapid Palatal Expansion) technique resulted in transverse skeletal expansion without the undesired dentoalveolar compensations or drawbacks. It also resulted in widening of the nasal cavity and zygomatic bone. ALT-RAMEC (Alternate Rapid Maxillary Expansion and Constriction) in literature proved to be advantageous over conventional RME in producing subluxation and sutural displacement to facilitate maxillary protraction in skeletal class III growing patients.The current study investigates the efficacy of a combination of MARPE/ ALT-RAMEC techniques to expand the maxilla in adult cases of transverse maxillary deficiency. It compares the proportion of success cases in patients who are treated with MARPE/ ALT-RAMEC to those treated using MARPE (conventional). It also describes the circum-maxillary sutural displacement in patients treated with both techniques, it hypothesizes that it will result in transverse skeletal expansion as well as sutural subluxation and displacement in young adult ages, which may be a sign of hope in the treatment of antero-posterior deficiency in adults without resorting to surgery. It also will describe the dento-skeletal changes (the amount of dental tipping) and the respiratory changes that occurred after applying the two different expansion techniques. It will also compare clinically, the changes occur gingivally (Gingival recession and Pocket depths) between pre-treatment and post-expansion periods.

DETAILED DESCRIPTION:
Patient with functional or esthetic complain (malocclusion) attending Dental Clinics in Al-Azhar University seeking orthodontic treatment, will be screened. Orthodontic young adult patients with transverse maxillary deficiency (as a primary diagnosis) will be selected from the list (by the study operator), based on inclusion and exclusion criteria. For this research purpose all subjects, whatever their number, who met the inclusion criteria, will be informed details of the expansion procedure, and about the whole study purposes, risks and benefits. Patient who agree to be a part of this research work, informed written consent will be taken from them. The patient will be divided randomly into two studying group, with a control group, Group A: (MARPE/ Conven), who will receive MARPE with its conventional expansion, and interventional group, Group B: who will receive a combination of MARPE/ALT-RAMEC technique. This randomization process will be carried out by the study operator using 30 sealed and shuffled envelopes, to blind both the operator and the participants during assignment to the groups. When a patient selects a group name, the operator will enroll him/her in the specific group list with allocation ratio 1:1 (15 patients in each group). Patient first visit (after assignment in the study) will take about 1 hour for preliminary evaluation, and T1 CBCT imaging. extra and intra oral assessment will be carried out to assess the dentition, occlusion type, periodontal status, and oral hygiene. Pretreatment CBCT imaging, gingival recession depths, and sulcus depths, will be taken as T1 records and interdental separating elastics will be used mesial and distal to 1st molars to provide adequate space for 1st molar banding.

Then a second visit will be required for impression taking, where orthodontic 1st molar bands will be selected and fitted properly in position for conventional alginate transfere impression to be taken for appliance laboratory construction. After that, dental separators will be reinserted again in their position. After which, and during the third visit (which might be the longest, 2 hours visit) the appliance will be loaded intraorally after local anesthesia infiltration using 4 mini-screws with previously planned length according to each patient palatal bone and soft tissue height. Then immediate activations (2-3 initial quarter turns), written hygiene, and activation instructions will be given to the patients in each group. In Group A (MARPE/conven) (Control), patients will open 2 quarter turn (0.2 mm) in the morning, and 2 quarter turn in the evening until overcorrection achieved. While in Group B (MARPE/ALT-RAMEC) (Interventional), patients will open 2 quarter turn (0.2mm) in the morning, and 2 in the evening in the first week, then alternate with closing 2 quarter turn in the morning and 2 in the evening in the second week. And then continuing opening and closing till end with opening in the 7th week and continue opening until overcorrection achieved. Patients will be followed up every week (1/2 an hour visit) for assessment of oral hygiene and interdental diastema appearance. In control group, if patients showed central diastema before 2-3 week , they will continue expansion till achieving overcorrection. But if they didn't show diastema after the 2-3 weeks, they will be terminated from the study and referred to maxillofacial surgery department for surgically assisted rapid palatal expansion (SARPE). In MARPE/ALT-RAMEC group, if patients showed diastema before 7-8 weeks of alternating expansion and constriction, they will continue only expansion till achieving overcorrection. But if they didn't; they will be terminated from the study and referred to maxillofacial surgery department for SARPE. All patients at the end of their expansion protocol, will get their T2 CBCT imaging and intra- oral measurements. Data collection from T1 and T2 CBCT records will be done by the study operator and then will be repeated again after 2 weeks of complete data collection by the same operator for data reliability. The patients who continue the expansion will be followed up until overcorrection is achieved which would take about 1-2 weeks after confirmation of median diastema event. The overall duration of participant involvement in group A (Control) is about 3-4 weeks, while in group B (Interventional) it will range from 8- 9 weeks.

ELIGIBILITY:
Inclusion Criteria:

* All cases showed maxillary skeletal deficiency. (Antero-posterior, or Transverse unilateral/ bilateral posterior cross bite).
* No history of facial orthopedic or orthognathic treatment before.
* No craniofacial anomaly or had history of serious craniofacial injuries.
* No history of serious medical illness such as (heart conditions, organ transplants, immune-compromised health issues, or cancer in patients undergoing chemotherapy or radiation treatments) or chronic diseases such as (Diabetes mellitus). As they are patients highly susceptible to infection which may result in worsening their medical status or even in a fatality in case of absence or inadequacy of precautions and proper pre/post medication coverage.
* Good oral hygiene and non-smoking habit.

Exclusion Criteria:

* Patient with missing or impacted 1st molars
* Patients with chronic gingival inflammation, gingival recession, or bone resorption.
* High gag reflex patients

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Transverse palatal Expansion | 2-9 weeks
  Achieving skeletal expansion in the posterior cross bite, which will be observed clinically by mid-palatal suture splitting (central diastema) then molar overcorrection, when the palatal cusp of either maxillary first molar came in contact with the corresponding buccal cusp tips of the mandibular first molar.
Sutural Displacement | 2-9 weeks
  Producing increased circum-maxillary sutural displacement measured from CBCT images, when comparing MARPE with ALT-RAMEC than MARPE with its conventional use.

CONTACTS AND LOCATIONS:
Overall Officials: Norma Ab Rahman, Study Director — Universiti Sains Malaysia
Locations (1):
- Universiti Sains Malaysia, Kubang Kerian, Kelantan, Malaysia

REFERENCES:
- [Derived] Allam A, Mostafa M, Ahmad B, Salama A, Rahman NA. The sutural and dentoskeletal effects of alternate expansion and constriction of deficient maxilla in young adults: a randomized controlled clinical trial. BMC Oral Health. 2025 Jul 13;25(1):1156. doi: 10.1186/s12903-025-06489-y. PMID 40653475